CLINICAL TRIAL: NCT02733107
Title: The Efficacy and Safety of Apatinib Combined With Etoposide in Advanced Non-small Cell Lung Cancer Patients Failed to Previous at Least 2rd Line Treatments
Brief Title: The Efficacy and Safety of Apatinib Combined With Etoposide in Heavily Pretreated Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xueqin Yang, PHD, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACEL
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Apatinib; Etoposide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib+Etoposide (Other): Apatinib combined with Etoposide
  Interventions: Drug: Apatinib; Drug: Etoposide

INTERVENTIONS:
Drug: Apatinib — Apatinib, 250mg daily, po, continue until disease progression
Drug: Etoposide — Etoposide, 50mg daily, po, day 1 to day 20, repeat Q 4 weeks until disease progression
  Other Names: VP-16

SUMMARY:
The development of anti-angiogenesis drugs has led to renewed enthusiasm in lung cancer treatments. Apatinib is a tyrosine kinase inhibitor which selectively inhibits the vascular endothelial growth factor receptor-2 (VEGFR-2). Etoposide is an oral preparation for lung cancer which is recommended by NCCN guideline. The investigators wondered whether these two drugs have synergistic effects when treating advanced non-small cell lung cancer patients who failed to previous at least 2nd line treatments. Thus, the aim of this trial is to investigate the efficacy and safety of apatinib combined with etoposide in heavily pretreated advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Obtain of informed consent.
* Histologically or cytologically confirmed non-small cell lung cancer.
* World Health Organization (WHO) performance status (PS) of 0 to 2.
* Measurable lesions as defined by RECIST criteria.
* Second-line or more treatments.
* Wild type of epidermal-growth-factor receptor (EGFR).
* Life expectancy ≥12 weeks.
* Organ functions normal, as defined below, within two weeks of randomization:

  • Hb≥90g/L Absolute neutrophils count(ANC)≥1.5×109/L Platelets≥80×109/L Serum bilirubin≤2×ULN; Aspartate transaminase(AST) and alanine transaminase (ALT)≤2.5×ULN(≤5×ULN if liver metastases) Creatinine clearance≥45ml/min or Cr≤1.25×ULN.
* Females of child-bearing potential must have negative serum pregnancy test.
* Sexually active males and females (of childbearing potential) willing to practice contraception during the study.

Exclusion Criteria:

* Small cell lung cancer.
* Newly diagnosed Central Nervous System (CNS) metastases that have not yet been definitively treated with surgery and/or radiation.
* Uncontrolled hypertension.
* Myocardial ischemia or infarction more than stage II, cardiac insufficiency.
* Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy.
* Difficulties in taking pills (inability to swallow tablets,GI tract resection, chronic bacillary diarrhea and intestinal obstruction).
* Hemoptysis, more than 2.5ml daily.
* Thrombosis in 12 months, including pulmonary thrombosis, stoke, or deep venous thrombosis.
* Unhealed bone fracture or wound for long time.
* Received big surgery, had bone fracture or ulcer in 4 weeks.
* Urine protein≥++, or urine protein in 24 hours≥1.0g.
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | evaluated in 24 months since the treatment began
  the first day of treatment to the date that disease progression is reported

SECONDARY OUTCOMES:
Objective Response Rate | tumor assessment every 6-8 weeks since the treatment began，up to 24 months
  the ratio between the number of responders and number of patients assessable for tumor response
Overall survival | the first day of treatment to death or last survival confirm date,up to 24 months
Side effects | evaluated in the 24th month since the treatment began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou C, Wu YL, Chen G, Liu X, Zhu Y, Lu S, Feng J, He J, Han B, Wang J, Jiang G, Hu C, Zhang H, Cheng G, Song X, Lu Y, Pan H, Zheng W, Yin AY. BEYOND: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Study of First-Line Carboplatin/Paclitaxel Plus Bevacizumab or Placebo in Chinese Patients With Advanced or Recurrent Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Jul 1;33(19):2197-204. doi: 10.1200/JCO.2014.59.4424. Epub 2015 May 26. PMID 26014294
- [Result] Okamoto I, Miyazaki M, Takeda M, Terashima M, Azuma K, Hayashi H, Kaneda H, Kurata T, Tsurutani J, Seto T, Hirai F, Konishi K, Sarashina A, Yagi N, Kaiser R, Nakagawa K. Tolerability of nintedanib (BIBF 1120) in combination with docetaxel: a phase 1 study in Japanese patients with previously treated non-small-cell lung cancer. J Thorac Oncol. 2015 Feb;10(2):346-52. doi: 10.1097/JTO.0000000000000395. PMID 25299232